CLINICAL TRIAL: NCT05024994
Title: A Phase II Clinical Trial of E7820 for Patients With Relapsed/Refractory Myeloid Malignancies With Mutations in Splicing Factor Genes.
Brief Title: A Study of E7820 in People With Bone Marrow (Myeloid) Cancers
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Memorial Sloan Kettering Cancer Center (Other)
Collaborators: Eisai Inc. (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 21-159
Record Dates: First submitted 2021-08-23; First posted 2021-08-27 (Actual); Last update posted 2025-06-22 (Actual); Status verified 2025-06

CONDITIONS: Acute Myeloid Leukemia; Myelodysplastic Syndromes; Chronic Myelomonocytic Leukemia
Keywords: E7820; Bone Marrow cancers; Myeloid; Relapsed/Refractory; Mutations in Splicing Factor Genes; 21-159
MeSH Terms: conditions — Leukemia, Myeloid, Acute; Myelodysplastic Syndromes; Leukemia, Myelomonocytic, Chronic; Recurrence | interventions — N-(3-cyano-4-methyl-1H-indol-7-yl)-3-cyanobenzene-sulfonamide

STUDY DESIGN:
Intervention Model Description: This is a phase II study exploring the efficacy of E7820 in patients with relapsed and refractory myeloid malignancies with mutations in splicing factors.
Oversight: FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (1):
- E7820 (Experimental): Each patient will receive daily administration of E7820. The starting dose for every patient will be 100 mg daily but the dose can subsequently be reduced if excessive toxicity is encountered.
  Interventions: Drug: E7820

INTERVENTIONS:
Drug: E7820 — 100mg of E7820 QD

SUMMARY:
The researchers are doing this study to find out whether E7820 is an effective treatment for people with relapsed/refractory myeloid cancers with mutations in splicing factor genes. Participants will have acute myeloid leukemia (AML), myelodysplastic syndromes (MDS), or chronic myelomonocytic leukemia (CMML).

ELIGIBILITY:
Inclusion Criteria:

1. Subject is ≥ 18 years of age at the time of signing informed consent 2. Subject is willing and able to adhere to the study visit schedule and other protocol requirements. 3. Subject has relapsed or refractory MDS, AML or CMML with a previously defined hotspot splicing factor mutation in SF3B1, SRSF2, U2AF1, or U2AF2 (with hotspot mutations as defined by OncoKB) or a nonsense or frameshift mutation in ZRSR2. A splicing factor mutation is required to be detected on next generation sequencing from bone marrow aspirate or peripheral blood at any timepoint within the 6 months prior to screening for the study.

a. Relapsed AML is defined as: i. The appearance of 5% or greater myeloblasts in the bone marrow or peripheral blood after achieving a CR (MRD positive or negative), CRh, or CRi

1. Patients with mutations in FLT3, IDH1 or IDH2 must have failed or been intolerant of an FDA approved FLT3, IDH1 or IDH2 inhibitor before enrolling on study.

b. Refractory AML is defined as failure to achieve a CR, CRh, or CRi after one of the following regimens: i. Two cycles of intensive induction chemotherapy with a cytarabine containing regimen (e.g. 7+3, MEC, HIDAC, etc.) ii. Two cycles of HMA/venetoclax or LDAC/glasdegib iii. 4 cycles of HMA monotherapy c. Relapsed MDS is defined as: i. Any relapse after achieving an IWG defined response. d. Refractory MDS is defined as: i. For patients with intermediate, high or very high risk disease by IPSS-R, the failure to achieve a response (as per IWG 2006 criteria) after 4 cycles of HMA monotherapy or 2 cycles of HMA + venetoclax.

ii. For patients with very low and low risk disease by IPSS-R failure to achieve hematologic improvement or loss of hematologic improvement after treatment with standard of care agents such as ESAs, Luspatercept (for MDS with ringed sideroblasts) and lenalidomide (for pts with a 5q-).

e. Relapsed CMML is defined as: i. Any relapse after achieving an IWG defined response. f. Refractory CMML is defined as: i. Failure to achieve a response (as per IWG 2006 criteria) after 4 cycles of HMA monotherapy or 2 cycles of HMA + venetoclax.

4. Subject has an Eastern Cooperative Oncology Group (ECOG) performance status of 0-3 5. Subject has adequate organ function defined as:

1. Serum aspartate aminotransferase/serum glutamic oxaloacetic transaminase (AST/SGOT) and alanine aminotransferase (ALT/SGPT) ≤ 3 x ULN, unless considered due to organ involvement by the patient's myeloid malignancy (in that case a cut off of ≤ 5 x ULN will be used)
2. Serum direct bilirubin < 1.5 x ULN.
3. Creatinine clearance ≥ 60 mL/min based on the Cockroft-Gault glomerular filtration rate (GFR) estimation.
4. Females of childbearing potential may participate provided they have a negative serum pregnancy test at screening and a negative serum OR urine pregnancy test within 72 hours of starting on treatment. Females and male participants with female partners of childbearing potential also must agree to either abstain from sexual intercourse or use a highly effective method of contraception while on study and for 4 months after completing the study treatment.

   6. There are no limits on transfusion and/or growth factor support for enrollment.

   7. In case of leukemic organ involvement, patients with creatinine clearance > 30 ml/min and bilirubin ≤ 2.0 x ULN will be eligible to be included.

   Exclusion Criteria:
   1. Patients with acute promyelocytic leukemia
   2. Subject has immediate life-threatening, severe complications of their myeloid malignancy such as uncontrolled bleeding, pneumonia with hypoxia or shock, and/or disseminated intravascular coagulation
   3. Subject has significant active cardiac disease within 6 months prior to the start of study treatment, including New York Heart Association (NYHA) class III or IV congestive heart failure; acute coronary syndrome (ACS); and/or stroke or left ventricular ejection fraction (LVEF) <40% by echocardiogram (ECHO) or multi-gated acquisition (MUGA) scan obtained within 28 days prior to the start of study treatment.
   4. Subject has active viral infection with human immunodeficiency virus (HIV), or active infection with hepatitis B virus (HBV) or hepatitis C virus (HCV). Patients with HIV that is controlled with HAART are eligible to participate.
   5. Subject is known to have dysphagia, short-gut syndrome, gastroparesis, or other conditions that limit the ingestion or gastrointestinal absorption of drugs administered orally.
   6. Subject has active uncontrolled systemic fungal, bacterial, or viral infection (defined as ongoing signs/symptoms related to the infection without improvement despite appropriate antibiotics, antiviral therapy, and/or other treatment).
   7. Subject has QTc interval (i.e., Fridericia's correction [QTcF]) ≥ 480 ms or other factors that increase the risk of QT prolongation or arrhythmic events (e.g., heart failure family history of long QT interval syndrome) at screening. Patients with left bundle branch block or right bundle branch block with prolonged QTc will be allowed to enroll on the trial with medical monitor approval.
   8. Female subject who is pregnant or lactating.
   9. Subject with known hypersensitivity to sulfa medications

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 12 (Actual)
Dates: Start 2021-08-13 (Actual); Primary Completion 2025-06-19 (Actual); Study Completion 2025-06-19 (Actual)

PRIMARY OUTCOMES:
response rate | 1 year
  Response to treatment and treatment decisions in all participants will be determined based on the 2017 ELN criteria for AML 2 and the International Working Group 2006 criteria for MDS 3 and 2015 for CMML4.

CONTACTS AND LOCATIONS:
Overall Officials: Eytan Stein, MD, Principal Investigator — Memorial Sloan Kettering Cancer Center
Locations (7):
- United States (7):
  - University of Miami (Data Collection AND Specimen Analysis Only), Miami, Florida
  - Memorial Sloan Kettering Basking Ridge, Basking Ridge, New Jersey
  - Memorial Sloan Kettering Monmouth, Middletown, New Jersey
  - Memorial Sloan Kettering Bergen, Montvale, New Jersey
  - Memorial Sloan Kettering Commack, Commack, New York
  - Memorial Sloan Kettering Westchester (All protocol activities), Harrison, New York
  - Memorial Sloan Kettering Nassau, Uniondale, New York

IPD SHARING:
Plan to Share IPD: Yes
Memorial Sloan Kettering Cancer Center supports the international committee of medical journal editors (ICMJE) and the ethical obligation of responsible sharing of data from clinical trials. The protocol summary, a statistical summary, and informed consent form will be made available on clinicaltrials.gov when required as a condition of Federal awards, other agreements supporting the research and/or as otherwise required. Requests for deidentified individual participant data can be made beginning 12 months after publication and for up to 36 months post publication. Deidentified individual participant data reported in the manuscript will be shared under the terms of a Data Use Agreement and may only be used for approved proposals. Requests may be made to: crdatashare@mskcc.org.

REFERENCES:
- [Derived] Bewersdorf JP, Stahl M, Taylor J, Mi X, Chandhok NS, Watts J, Derkach A, Wysocki M, Lu SX, Bourcier J, Hogg SJ, Rahman J, Chaudhry S, Totiger TM, Abdel-Wahab O, Stein EM. E7820, an anti-cancer sulfonamide, degrades RBM39 in patients with splicing factor mutant myeloid malignancies: a phase II clinical trial. Leukemia. 2023 Dec;37(12):2512-2516. doi: 10.1038/s41375-023-02050-4. Epub 2023 Oct 9. No abstract available. PMID 37814121
- See also: Memorial Sloan Kettering Cancer Center — http://www.mskcc.org/mskcc/html/44.cfm